CLINICAL TRIAL: NCT02004197
Title: Phytomedicine-based and Quadruple Therapies in Helicobacter Pylori Infection. A Comparative Randomized Trial
Brief Title: Quadruple and Phytomedicine-based Therapies in H. Pylori Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hafiz Muhammad Asif (Other)
Responsible Party: Sponsor-Investigator, Hafiz Muhammad Asif, Doctor, Shifa Ul Mulk Memorial Hospital
Organization: Shifa Ul Mulk Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Asif-HP-001
Record Dates: First submitted 2013-08-20; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Helicobacter Pylori [H. Pylori] as the Cause of Diseases
MeSH Terms: interventions — Omeprazole; Amoxicillin; ranitidine bismuth citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pylorex plus (Experimental): Pylorex plus consisting of medicinal plants.
  Interventions: Drug: Quadruple Allopathic therapy; Drug: Pylorex plus
- Quadruple therapy (Active Comparator): Omeprazole, Amoxicillin, Metronodazole and TRITEC (ranitidine bismuth citrate)
  Interventions: Drug: Quadruple Allopathic therapy; Drug: Pylorex plus

INTERVENTIONS:
Drug: Quadruple Allopathic therapy
  Other Names: Omeprazol; Amoxicillin; Metronodazole; TRITEC (ranitidine bismuth citrate)
Drug: Pylorex plus

SUMMARY:
Helicobacter pylori is strongly associated to the development of gastrointestinal disorders. Emerging antibiotic resistance and poor patient compliance of modern therapies has resulted in significant eradication failure. Clinical trial was conducted to see the efficacy of current quadruple and phytomedicine-based therapies for the eradication of H. pylori infection and relief in its associated symptoms in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

1. The patients suffering from H. pylori infection
2. Patients having no previous record of treatment against H. pylori infection
3. Patients living in Karachi, Rawalpindi and Bahawalpur
4. Patients having no pathological complications on routine examination
5. All socioeconomic classes were included in the study
6. Male and female patients between 15 to 45 years of age

Exclusion Criteria:

1. there was peptic ulceration, gastrointestinal bleeding or gastric carcinoma
2. if history of use of antibiotics, proton-pump inhibitors or bismuth compound in the last one month before test
3. any patient found to be allergic or intolerant to therapeutic regimens
4. they failed to report for follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate was the primary endpoint, which was considered to be achieved on the basis of a negative urea breath and stool antigen test four weeks after the end of treatment | 1 month

SECONDARY OUTCOMES:
The secondary endpoint was the improvement in the clinical features as assessed by an improvement in dyspepsia scores | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Khan Usman Ghani, Ph. D, Study Director — Hamdard University Karachi
Locations (2):
- Pakistan (2):
  - clinical trial was conducted in high risk areas of Pakistan such as Karachi, Bahawalpur, Islamabad and Rawalpindi at Shifa-Ul-Mulk Memorial Hospital, Hamdrad University Karachi, Bahawalpur Victoria Hospital and Nawaz Salik Hospital respectively, Karachi
  - Shifa Ul MUlk Memorial Hospital, Karachi